CLINICAL TRIAL: NCT05619666
Title: Acute Rehabilitation in Patients With COVID-19 Pneumonia a Single Center Experience From a Developing Country
Brief Title: Acute Rehabilitation in Patients With COVID-19 Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut za Rehabilitaciju Sokobanjska Beograd (Other)
Responsible Party: Principal Investigator, Tamara Filipovic, Teaching assistant, Institut za Rehabilitaciju Sokobanjska Beograd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02/269-1
Record Dates: First submitted 2022-11-14; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Rehabilitation; Physical Medicine
Keywords: Acute rehabilitation; COVID-19 pneumonia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severity of COVID-19 infection (Other): Based on the severity of Covid-19 infection patients were divided into 2 groups: First group (MMG) mild to moderate group and second group (SSG) stable severe group.
  Interventions: Procedure: Acute rehabilitation program

INTERVENTIONS:
Procedure: Acute rehabilitation program — Patients included in the study started the rehabilitation program when they were hemodynamic stable, when it was determined that it was safe for patients. Until discharge from the hospital, a re-evaluation of neuromuscular and respiratory function was performed.

SUMMARY:
COVID-19 can have different clinical manifestations including myalgia, arthralgia, neurological, cardiac, psychological and other manifestations.These patients are at greater risk of developing consequences of prolonged bed rest. Therefore physical medicine and rehabilitation could have an important role in the multidisciplinary treatment of these issues. Early respiratory and neuromuscular rehabilitation is necessary to improve functional physical limitations, performance, muscle strength, endurance as well as cognitive and emotional domains. Some studies proposed that rehabilitation protocols in the inpatient setting include early mobilisation, strength and endurance training with the aim of reducing weakness and dependency. This Study aimed to detect the effects of rehabilitation in patients with Covid-19 who were admitted in temporary Covid hospital in Serbia. Furthermore, to emphasize the importance of functional assessment of the patients, in identifying their problems and selections of priorities in planning the best therapeutic protocol.

ELIGIBILITY:
Inclusion Criteria:

* Positive pharyngeal or nasal swab for SARS CoV-2, 3) SP O2> 94% on admission, 4) body temperature under 37.5 5) Clinical stability defined by ability to perform bedside active mobilization without a reduction of oxygen saturation (SpO2) below 92%;

Exclusion Criteria:

* 1) SP o2 < 94% on admission, 2) Moderate and severe heart failure (grade III and IV, NY heart Association), 3) Paresis or plegia as a result of CVI or neurodegenerative disease, 4) Impaired cognitive status.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
functional outcome of activity of daily living | up to three weeks
  Bartel index (BI)
functional outcome of cardiovascular and respiratory system | up to three weeks
  six minute walk test (6MWT)
functional outcome for assesing dyspnea | up to three weeks
  Borg scale for dyspnea,
functional outcome of mobility | up to three weeks
  "Time Up and Go" test (TUG)
functional outcome of lower limbs strength | up to three weeks
  "Sit To Stand" test (STS)
functional outcome of static balance | up to three weeks
  "One Leg Stance Test" (OLST)

CONTACTS AND LOCATIONS:
Locations (2):
- Serbia (2):
  - Tamara Filipovic, Belgrade
  - Institute for Rehabilitation, Belgrade